CLINICAL TRIAL: NCT00000791
Title: A Phase II Double-Blind Study of Two Doses of SC-49483 in Combination With Zidovudine (ZDV) Versus ZDV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: G D Searle (Industry); Glaxo Wellcome (Industry)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 259; 11236 (Registry Identifier: DAIDS-ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Antiviral Agents; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — glycovir; Zidovudine

INTERVENTIONS:
Drug: Glycovir
Drug: Zidovudine

SUMMARY:
To determine the safety and anti-HIV activity of two doses of SC-49483 in combination with zidovudine (AZT) versus AZT alone. To determine the influences of viral phenotype on the anti-HIV activity of these treatment regimens.

SC-49483 has no inherent activity against HIV-1 but is converted in the intestinal wall to SC-48334, which has demonstrated anti-HIV activity. Since SC-49483 causes significantly less gastrointestinal toxicity than SC-48334, the combination of SC-49483 with AZT may improve the benefits of both drugs in patients with HIV infection.

DETAILED DESCRIPTION:
SC-49483 has no inherent activity against HIV-1 but is converted in the intestinal wall to SC-48334, which has demonstrated anti-HIV activity. Since SC-49483 causes significantly less gastrointestinal toxicity than SC-48334, the combination of SC-49483 with AZT may improve the benefits of both drugs in patients with HIV infection.

Patients are randomized to receive AZT alone or in combination with one of two doses of SC-49483, administered three times daily. Treatment continues for 16 to 24 weeks. Per 07/19/94 amendment: At the end of 24 weeks, blinded treatment continues for an additional 4 weeks, at which time patients may receive open-label drug on an optional basis for 90 days.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Required:

* PCP prophylaxis (trimethoprim/sulfamethoxazole, dapsone, or aerosolized pentamidine) in patients with CD4 count <= 200 cells/mm3.

Allowed:

* Topical antifungal agents, ketoconazole, fluconazole, and itraconazole for candidiasis or disseminated fungal infections, as medically indicated.
* Maintenance therapy for Mycobacteria disease with isoniazid, ethambutol, rifampin, pyrazinamide, clofazimine, ciprofloxacin, clarithromycin, or rifabutin.
* Maintenance therapy for toxoplasmosis with pyrimethamine, sulfadiazine, or clindamycin.
* Maintenance therapy for herpes simplex virus with acyclovir at <= 1000 mg/day.
* Recombinant erythropoietin and G-CSF, if indicated.
* Antibiotics for bacterial infections.
* Symptomatic treatment such as antipyretics, analgesics, nonsteroidal anti-inflammatory agents, and antiemetics.

Concurrent Treatment:

Allowed:

* Localized radiation therapy and limited intralesional therapy for cutaneous Kaposi's sarcoma.

Patients must have:

* Documented HIV infection.
* Per 07/19/94 amendment, one of the following:
* CD4 count 150 - 350 cells/mm3 within 60 days prior to study entry AND prior AZT for no more than 12 months cumulative (given with or without ddI or ddC).
* CD4 count 50 - 350 cells/mm3 within 60 days prior to study entry AND no prior antiretroviral therapy.
* MT-2 cell assay within 60 days prior to study entry.

NOTE:

* Minimal Kaposi's sarcoma is permitted.

Exclusion Criteria

Co-existing Condition:

Patients with the following condition are excluded:

* Malignancy other than minimal Kaposi's sarcoma.

Concurrent Medication:

Excluded:

* Antiretroviral therapies (other than study drug).
* Biologic response modifiers.
* Systemic corticosteroids for > 21 consecutive days.
* Foscarnet.
* Systemic cytotoxic chemotherapy for a malignancy.

Patients with the following prior conditions are excluded:

* History of cataracts.
* History of intolerance to AZT at <= 600 mg/day.
* Unexplained temperature >= 38.5 degrees C that persists for any 7 days within the 30 days prior to study entry.
* Chronic diarrhea (defined as >= 3 stools per day) that persists for any 15 days within the 30 days prior to study entry.

Prior Medication:

Excluded:

* More than 6 months (more than 12 months per 07/19/94 amendment) cumulative prior therapy with AZT.
* Prior induction or maintenance therapy with foscarnet.
* Any investigational drug within 30 days prior to study entry.
* Prior SC-49483 or SC-48334.
* Prior ddC, ddI, or stavudine (d4T) as monotherapy.
* Interferon or interleukin within 30 days prior to study entry.
* Prior non-nucleoside reverse transcriptase inhibitors (e.g., NVP, ATV).
* Systemic corticosteroids for > 21 consecutive days.
* Acute treatment for a serious infection or any opportunistic infection within 14 days prior to study entry.
* Prior combination therapy with AZT, ddI, and/or ddC within 30 days prior to study entry.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210
Dates: Study Completion 1995-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fischl MA, Study Chair; Saag M, Study Chair
Locations (22):
- United States (22):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - USC CRS, Los Angeles, California
  - Stanford CRS, Palo Alto, California
  - Ucsf Aids Crs, San Francisco, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Northwestern University CRS, Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Weiss Memorial Hosp., Chicago, Illinois
  - Cook County Hosp. CORE Ctr., Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Methodist Hosp. of Indiana, Indianapolis, Indiana
  - St. Louis ConnectCare, Infectious Diseases Clinic, St Louis, Missouri
  - Washington U CRS, St Louis, Missouri
  - SUNY - Buffalo, Erie County Medical Ctr., Buffalo, New York
  - Beth Israel Med. Ctr. (Mt. Sinai), New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Wake County Health and Human Services CRS, Raleigh, North Carolina
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
  - University of Washington AIDS CRS, Seattle, Washington

REFERENCES:
- [Background] Johnson VA, Bassett RL, Stanley KE, Saag MS, Fischl MA. Predictors of syncytium-inducing viral phenotype in a phase II double-blind trial of SC-49483 plus ZDV vs. ZDV. Conf Retroviruses Opportunistic Infect. 1997 Jan 22-26;4th:102 (abstract no 205)